CLINICAL TRIAL: NCT00077129
Title: Phase II Trial Of Paclitaxel Plus Carboplatin In Patients With Metastatic Or Locally Advanced Collecting Duct Renal Cell Cancer
Brief Title: Paclitaxel and Carboplatin in Treating Patients With Locally Advanced or Metastatic Renal Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Group Chair, Eastern Cooperative Oncology Group
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000349502; E2803
Record Dates: First submitted 2004-02-10; First posted 2004-02-11 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Kidney Cancer
Keywords: stage III renal cell cancer; stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: carboplatin
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Giving more than one drug may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving paclitaxel together with carboplatin works in treating patients with locally advanced or metastatic collecting duct renal cell cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in patients with locally advanced or metastatic collecting duct renal cell cancer treated with paclitaxel and carboplatin.

Secondary

* Determine the tolerability of this regimen in these patients.

OUTLINE: This is an open-label, multicenter study.

Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of unacceptable toxicity or disease progression.

Patients are followed every 3 months for 2 years and then every 6 months for 1 year.

PROJECTED ACCRUAL: A total of 14-22 patients will be accrued for this study within 4.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed collecting duct renal cell carcinoma

  * Advanced locally recurrent or metastatic disease
  * Not amenable to resection
* Measurable disease
* No active CNS metastases

  * Patients with CNS metastases previously treated with surgical resection and/or radiotherapy are eligible provided there is no evidence of disease progression by head CT scan or MRI at 3 months after the completion of definitive therapy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* WBC ≥ 3,000/mm^3
* Absolute granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN

Renal

* Creatinine ≤ 2 times ULN

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No peripheral neuropathy greater than grade 1
* No other prior malignancy except for curatively treated cancer from which the patient has been disease-free for the length of time considered appropriate for cure of the specific cancer
* No known hypersensitivity to Cremophor EL
* No active serious infection
* No other serious underlying medical condition that would preclude study therapy
* No dementia or significantly altered mental status that would preclude giving informed consent

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No more than 2 prior biologic response modifier (BRM) regimens

  * Regimens may have included interleukin-2 and/or interferon alfa
* At least 4 weeks since prior BRM therapy

Chemotherapy

* Not specified

Endocrine therapy

* Concurrent corticosteroids allowed

Radiotherapy

* See Disease Characteristics
* Prior radiotherapy allowed provided there is measurable disease that has not been irradiated OR there is clear evidence of tumor progression in an irradiated site
* At least 4 weeks since prior radiotherapy
* No concurrent external beam radiotherapy

Surgery

* See Disease Characteristics
* No concurrent major surgery

Other

* No other concurrent anticancer drugs

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2006-06-01 (Actual); Primary Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with clinical response

SECONDARY OUTCOMES:
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: David F. McDermott, MD, Study Chair — Beth Israel Deaconess Medical Center; Michael B. Atkins, MD, Study Chair — Beth Israel Deaconess Medical Center
Locations (35):
- United States (35):
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - Mercy Hospital and Medical Center, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - Midwest Center for Hematology/Oncology, Joliet, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - North Shore Oncology and Hematology Associates, Limited - Libertyville, Libertyville, Illinois
  - Northwest Medical Specialist, PC, Niles, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - Hematology/Oncology of the North Shore at Gross Point Medical Center, Skokie, Illinois
  - Midwest Cancer Research Group, Incorporated, Skokie, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - McFarland Clinic, P. C., Ames, Iowa
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - MeritCare Clinic - Bemidji, Bemidji, Minnesota
  - Our Lady of Mercy Medical Center Comprehensive Cancer Center, The Bronx, New York
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Medical Group, Fargo, North Dakota
  - St. Rita's Medical Center, Lima, Ohio
  - St. Luke's Hospital Cancer Center, Bethlehem, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin